CLINICAL TRIAL: NCT03098121
Title: Efficacy and Tolerability of Grazoprevir and Elbasvir in Peginterferon Alfa Plus Ribavirin Experienced Patients With Chronic Genotype 1 HCV and HIV Co-infection: a Non-randomised, Open-label Clinical Trial
Brief Title: Efficacy and Tolerability of Grazoprevir and Elbasvir in Patients With Chronic Genotype 1 HCV and HIV Co-infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYGH105034
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Genotype 1 HCV and HIV co-infection (Experimental): Patients with chronic Genotype 1 HCV and HIV co-infection, with or without resistance-associated substitution (RAS) of NS5A, received grazoprevir and elbasvir in a fixed-dose combination tablet once daily with ribavirin for 16 weeks, and patients with chronic genotype 1b received grazoprevir and elbasvir once daily for 12 weeks.
  Interventions: Drug: grazoprevir and elbasvir

INTERVENTIONS:
Drug: grazoprevir and elbasvir — For patients with chronic genotype 1a, with or without resistance associated variant (RAV) of NS5A, are expected to receive grazoprevir and elbasvir in a fixed-dose combination tablet once daily with ribavirin for 16 weeks, and for patients with chronic genotype 1b are expected to receive grazoprevir and elbasvir in a fixed-dose combination tablet once daily for 12 weeks.

SUMMARY:
This clinical study will evaluate whether grazoprevir and elbasvir is efficacious, safe, and well-tolerated in peginterferon alfa plus ribavirin experienced patients who inject drugs (PWID) and men who sex with men (MSM) with genotype 1 HCV and HIV co-infection.

DETAILED DESCRIPTION:
Primary Objective •To assess the efficacy of grazoprevir 100mg and elbasvir 50mg by determining the proportion of sustained virological response 12 weeks after the end of therapy (SVR12; HCV RNA concentration less than 10 IU/ mL at follow-up week 12) in peginterferon alfa plus ribavirin experienced patients with genotype 1 HCV and HIV co-infection, compared with treatment-naïve patients with 1 HCV and HIV co-infection.

Secondary Objective

•To assess the tolerability of grazoprevir 100mg and elbasvir 50mg in peginterferon alfa plus ribavirin experienced patients by measuring frequency of SAEs and AEs leading to discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women, at least 20 years of age with chronic genotype 1 HCV and HIV co-infection.
* HCV RNA > 10,000 IU/mL
* Stable antiretroviral therapy (ARV) with confirmed plasma HIV-1 RNA < 200 copies/mL
* CD4 T-cell count > 100 cells/L
* peginterferon alfa plus ribavirin failure: null response <1 log10 IU/mL reduction in HCV RNA at week 4; detectable HCV RNA since week 12 to the end of treatment; detectable HCV RNA for 12 to 24 weeks after the end of treatment; or discontinuation of peginterferon alfa plus ribavirin due to grade 3 or grade 4 adverse effects at any moment.

Exclusion Criteria:

* Decompensated liver disease (presence or history of ascites, oesophageal or gastric variceal bleeding, hepatic encephalopathy, or other signs of advanced liver diseases)
* Liver cirrhosis with Child-Pugh class B or C, or with a Child-Turcotte-Pugh score of more than 6 points and albumin below 3 g/dL or platelet count below 75,000/ μL
* History of malignant disease, or evidence of hepatocellular carcinoma
* ARV with protease inhibitor containing regimen HBsAg and HBV core antibody should be checked in all patients. HBsAg positive patients should be excluded from the study. HBV core antibody positive patients should be closely monitored for hepatitis flare or HBV reactivation during HCV treatment and post-treatment follow-up. Appropriate patient management should be instituted for HBV infection as clinically indicated.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 12 weeks after the end of therapy
  The proportion of sustained virological response 12 weeks after the end of therapy after the treatment of grazoprevir and elbasvir

SECONDARY OUTCOMES:
Severe adverse effects | during the treatment of grazoprevir and elbasvir
  The frequency of severe adverse effects leading to discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Yu Cheng, Principal Investigator — Taoyuan General Hospital
Locations (1):
- Taoyuan general hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The study will be conducted at 3 different hospitals, and the investigators will share the data with other researchers every 3 months
Supporting Information: Study Protocol
Time Frame: The data will become available in March 2019.
Access Criteria: The investigators will share the data and outcome via international conference

REFERENCES:
- [Background] Laguno M, Cifuentes C, Murillas J, Veloso S, Larrousse M, Payeras A, Bonet L, Vidal F, Milinkovic A, Bassa A, Villalonga C, Perez I, Tural C, Martinez-Rebollar M, Calvo M, Blanco JL, Martinez E, Sanchez-Tapias JM, Gatell JM, Mallolas J. Randomized trial comparing pegylated interferon alpha-2b versus pegylated interferon alpha-2a, both plus ribavirin, to treat chronic hepatitis C in human immunodeficiency virus patients. Hepatology. 2009 Jan;49(1):22-31. doi: 10.1002/hep.22598. PMID 19085908
- [Background] Chung RT, Andersen J, Volberding P, Robbins GK, Liu T, Sherman KE, Peters MG, Koziel MJ, Bhan AK, Alston B, Colquhoun D, Nevin T, Harb G, van der Horst C; AIDS Clinical Trials Group A5071 Study Team. Peginterferon Alfa-2a plus ribavirin versus interferon alfa-2a plus ribavirin for chronic hepatitis C in HIV-coinfected persons. N Engl J Med. 2004 Jul 29;351(5):451-9. doi: 10.1056/NEJMoa032653. PMID 15282352
- [Background] Torriani FJ, Rodriguez-Torres M, Rockstroh JK, Lissen E, Gonzalez-Garcia J, Lazzarin A, Carosi G, Sasadeusz J, Katlama C, Montaner J, Sette H Jr, Passe S, De Pamphilis J, Duff F, Schrenk UM, Dieterich DT; APRICOT Study Group. Peginterferon Alfa-2a plus ribavirin for chronic hepatitis C virus infection in HIV-infected patients. N Engl J Med. 2004 Jul 29;351(5):438-50. doi: 10.1056/NEJMoa040842. PMID 15282351
- [Background] Liu JY, Lin HH, Liu YC, Lee SS, Chen YL, Hung CC, Ko WC, Huang CK, Lai CH, Chen YS, Shih YL, Chung HC, Liang SH, Lin JN. Extremely high prevalence and genetic diversity of hepatitis C virus infection among HIV-infected injection drug users in Taiwan. Clin Infect Dis. 2008 Jun 1;46(11):1761-8. doi: 10.1086/587992. PMID 18433337
- [Background] Liu CH, Sheng WH, Sun HY, Hsieh SM, Lo YC, Liu CJ, Su TH, Yang HC, Liu WC, Chen PJ, Chen DS, Hung CC, Kao JH. Peginterferon plus Ribavirin for HIV-infected Patients with Treatment-Naive Acute or Chronic HCV Infection in Taiwan: A Prospective Cohort Study. Sci Rep. 2015 Nov 30;5:17410. doi: 10.1038/srep17410. PMID 26616669
- [Background] Naggie S, Cooper C, Saag M, Workowski K, Ruane P, Towner WJ, Marks K, Luetkemeyer A, Baden RP, Sax PE, Gane E, Santana-Bagur J, Stamm LM, Yang JC, German P, Dvory-Sobol H, Ni L, Pang PS, McHutchison JG, Stedman CA, Morales-Ramirez JO, Brau N, Jayaweera D, Colson AE, Tebas P, Wong DK, Dieterich D, Sulkowski M; ION-4 Investigators. Ledipasvir and Sofosbuvir for HCV in Patients Coinfected with HIV-1. N Engl J Med. 2015 Aug 20;373(8):705-13. doi: 10.1056/NEJMoa1501315. Epub 2015 Jul 21. PMID 26196665
- [Background] Wyles DL, Ruane PJ, Sulkowski MS, Dieterich D, Luetkemeyer A, Morgan TR, Sherman KE, Dretler R, Fishbein D, Gathe JC Jr, Henn S, Hinestrosa F, Huynh C, McDonald C, Mills A, Overton ET, Ramgopal M, Rashbaum B, Ray G, Scarsella A, Yozviak J, McPhee F, Liu Z, Hughes E, Yin PD, Noviello S, Ackerman P; ALLY-2 Investigators. Daclatasvir plus Sofosbuvir for HCV in Patients Coinfected with HIV-1. N Engl J Med. 2015 Aug 20;373(8):714-25. doi: 10.1056/NEJMoa1503153. Epub 2015 Jul 21. PMID 26196502
- [Background] Rockstroh JK, Nelson M, Katlama C, Lalezari J, Mallolas J, Bloch M, Matthews GV, Saag MS, Zamor PJ, Orkin C, Gress J, Klopfer S, Shaughnessy M, Wahl J, Nguyen BY, Barr E, Platt HL, Robertson MN, Sulkowski M. Efficacy and safety of grazoprevir (MK-5172) and elbasvir (MK-8742) in patients with hepatitis C virus and HIV co-infection (C-EDGE CO-INFECTION): a non-randomised, open-label trial. Lancet HIV. 2015 Aug;2(8):e319-27. doi: 10.1016/S2352-3018(15)00114-9. Epub 2015 Jul 9. PMID 26423374
- [Result] Bunchorntavakul C, Chavalitdhamrong D, Tanwandee T. Hepatitis C genotype 6: A concise review and response-guided therapy proposal. World J Hepatol. 2013 Sep 27;5(9):496-504. doi: 10.4254/wjh.v5.i9.496. PMID 24073301
- [Derived] Lin YC, Li SW, Ku SY, Hsieh HT, Lin MH, Chang SY, Wu WW, Sun NL, Cheng SH, Cheng CY. Grazoprevir/elbasvir in peginterferon alfa plus ribavirin experienced patients with chronic genotype 1 HCV/HIV co-infection: a non-randomized, open-label clinical trial. Infect Drug Resist. 2019 Apr 18;12:937-945. doi: 10.2147/IDR.S206938. eCollection 2019. PMID 31114268